CLINICAL TRIAL: NCT03715348
Title: A Pragmatic Pilot Randomised Phase II Controlled Trial of Prothrombin Complex Concentrates (PCC) Versus Fresh Frozen Plasma (FFP) in Adult Patients Who Are Undergoing Heart Surgery
Brief Title: Trial of PCC Versus FFP in Patients Undergoing Heart Surgery
Acronym: PROPHESY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 012507; 2018-003041-41 (EudraCT Number)
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2018-09

CONDITIONS: Bleeding; Surgery; Transfusion
Keywords: fresh frozen plasma; prothrombin complex concentrate; cardiac surgery
MeSH Terms: conditions — Hemorrhage; Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: Pragmatic pilot, open label, phase II randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Frozen Plasma (FFP) (Active Comparator): Patients randomised to the comparator arm will receive Fresh Frozen Plasma (FFP)
  FFP will be provide as a solution for intravenous administration, once thawed.
  The dose of the FFP will be ~ 15 mL/kg.
  Subjects may receive multiple doses of FFP as required if bleeding continues, as per usual care
  Interventions: Biological: Fresh Frozen Plasma
- Prothrombin Complex Concentrate (PCC) (Experimental): Patients randomised to the experimental arm will receive PCC at ~15 IU/kg. PCC will be reconstituted into a solution for intravenous administration.
  Subjects will receive a single dose of PCC, and if bleeding continues, standard treatment will be administered
  Interventions: Drug: Prothrombin Complex Concentrate (PCC)

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate (PCC) — PCC is a blood product produced through pooling of thousands of human plasmas, which is then treated to inactivate enveloped viruses. From the pooled plasma, vitamin K dependent clotting factors (factors II, VII, IX and X, and protein C and protein S), are selected to produce the concentrated form called PCC.
  Arms: Prothrombin Complex Concentrate (PCC)
Biological: Fresh Frozen Plasma — Fresh Frozen Plasma a blood component manufactured from whole blood collection.
  Arms: Fresh Frozen Plasma (FFP)

SUMMARY:
The PROPHESY trial is a single centre pilot trial investigating Fresh Frozen Plasma (FFP) or Prothrombin Complex Concentrate (PCC) treatment for patients who are bleeding during cardiac surgery, and who are NOT receiving a vitamin K antagonist agent (e.g. warfarin).

This pilot study will investigate the feasibility of delivering the different components of the trial, so that investigators can determine if it's feasible to move to a future large trial that will aim to compare the efficacy and safety of FFP versus PCC in adult patients who are actively bleeding during cardiac surgery.

DETAILED DESCRIPTION:
There are ~ 30,000 cardiac procedures performed each year in the United Kingdom (UK), and it is estimated that ~30% of these cases require plasma transfusion for management of bleeding during cardiovascular surgery. Bleeding after cardiac surgery that requires blood transfusion is associated with significant morbidity and mortality, resulting in substantial costs to the health service.

There have been no clinical trials that have compared the safety and efficacy of FFP versus PCC in cardiac surgery in patients who are bleeding, and who are not on vitamin K antagonists. In the UK, FFP transfusion is the standard treatment for management of bleeding: however, the use of PCC in this setting is rising, with several observational studies now demonstrating that it is safe, and that its administration is associated with reduced blood transfusion requirements, albeit no difference in other outcomes. Potential advantages of PCC over FFP are: increased concentration of clotting factors leading to faster improvement of reversing coagulopathy; improved ease and speed of administration; reduced fluid volume; and reduced incidence of immune modulatory side effects.

While observational studies have suggested that PCC can be safely administered in bleeding patients undergoing cardiac surgery, the clinical equipoise and, the lack of high quality evidence means that a randomised control trial is required to compare the clinical efficacy and safety of both in bleeding patients undergoing cardiac surgery not relating to warfarin. Prior to such a trial, the investigators will perform a single-centre pilot study to assess if individual components of a large trial are deliverable.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to give consent
* Any cardiovascular surgeries excluding procedures under exclusion criteria

Exclusion Criteria:

* Unable to consent
* Patients refusing blood transfusion for any reason
* First time isolated coronary artery bypass grafts (CABG)
* First time isolated aortic valve replacement (excluding active endocarditis)
* Thoraco-abdominal surgeries
* Minor surgeries that do not involve cardiopulmonary bypass
* Use of warfarin within four days
* Use of direct oral anticoagulants (i.e. dabigatran, rivaroxaban, apixaban or edoxaban) within 48 hrs (or 72 hours if patient has renal impairment - i.e. estimated glomerular filtration rate of <30ml/min)
* Inherited bleeding disorder (i.e. any inherited clotting factor deficiencies, or platelet disorders)
* Pregnancy
* Known or suspected allergy to FFP or PCC
* Known or suspected allergy to heparin, Sodium citrate dihydrate, sodium dihydrogenphosphate dihydrate and Glycine
* History of Heparin-induced thrombocytopenia
* Individuals who have Immunoglobulin A (IgA) deficiency with known antibodies against IgA
* Documented venous thromboembolism in the last three months
* Documented antiphospholipid syndrome
* Severe protein S deficiency
* Participation in another clinical trial, where the patient has received Investigational Medicinal Product in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Within 24 hours of surgery
  Proportion of eligible patients who consent to the study Proportion of patients who have consented and who bleed within 24 hours and who require FFP transfusion.

SECONDARY OUTCOMES:
Delivery of different components of the trial to see if a larger trial is feasible | Collected at 90 days or death, whichever occurs first
  The data collected from different trial componenets, such as study drugs administration, study procedure adherence and analysis of clinical outcome data will be combined and assessed to see whether it is feasible to successfully run this pilot as a larger, multi-centre trial
To compare the impact of FFP and PCC on the haemostatic capacity of bleeding patients after cardiac surgery | Within 24 hours of surgery
  Routine clotting tests and additional clotting tests will be performed to measure clotting factor levels, markers for clotting and anticoagulant activity in patients receiving FFP compare to PCC
Qualitative research involving completion of a Delphi survey to apprise the management and conduct of a larger trial | Completed over a 4 month period during the study follow-up stage
  Using the Delphi survey, information will be obtained from patient and public involvement (PPI) and healthcare professionals on the design/running of the larger trial, in order to understand how best to optimise identification and recruitment of participants, and to improve adherence to the trial procedures and protocol.
Qualitative research involving interviews of patients and healthcare professionals involved in PROPHESY to apprise the management and conduct of a larger trial | By the 90 days end of study visit
  Interviews will be conducted with 6 study subjects and 8 healthcare professionals involved in the PROPHESY trial to inform on the key aspects for the successful conduct and mangement of a larger trial

CONTACTS AND LOCATIONS:
Overall Officials: Laura Green, MBBS MsC MD(Res) MRCP FRCPath, Principal Investigator — Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Study results will be published in peer review journals and presented at national/international scientific meetings.
  The sponsor retains the right to review all publications prior to submission. Responsibility for ensuring accuracy of any publication from this study is delegated to the Chief Investigator.

REFERENCES:
- [Derived] Hayes K, Fernando MC, Jordan V. Prothrombin complex concentrate in cardiac surgery for the treatment of coagulopathic bleeding. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD013551. doi: 10.1002/14651858.CD013551.pub2. PMID 36408876
- [Derived] Green L, Roberts N, Cooper J, Field J, Gill R, Klein A, Agarwal S, Stanworth S, Johnston A, Monk V, O'Brien B. A pragmatic pilot phase II randomised controlled trial of prothrombin complex concentrates (PCC) versus fresh frozen plasma (FFP) in adult patients who are undergoing heart surgery (PROPHESY). Trials. 2019 Dec 9;20(1):684. doi: 10.1186/s13063-019-3759-8. PMID 31815658